CLINICAL TRIAL: NCT01949662
Title: A Preliminary Double-Blind Randomized Controlled Trial of Haloperidol and Lorazepam for Delirium in Patients With Advanced Cancer Admitted to a Palliative Care Unit
Brief Title: Haloperidol and Lorazepam for Delirium in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013-0345; NCI-2013-02351 (Registry Identifier: NCI CTRP); 1R21CA186000-01A1 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancers
Keywords: Advanced Malignant Solid Neoplasm; Delirium; Hematopoietic and Lymphoid Cell Neoplasm; Locally Advanced Malignant Solid Neoplasm; Malignant Solid Neoplasm; Neurotoxicity Syndrome; Questionnaires; Surveys; Acute palliative care unit
MeSH Terms: conditions — Delirium; Hematologic Neoplasms; Neurotoxicity Syndromes | interventions — Lorazepam; haloperidol decanoate; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorazepam + Haloperidol (Experimental): Participants given a single dose of lorazepam 3 mg by vein, in addition to a standardized dose of haloperidol 8 mg/day by vein, while in palliative care unit. Questionnaire completion at baseline, and every day while participant is in the palliative care unit. These questions will take about 20 minutes to complete
  Interventions: Drug: Lorazepam; Drug: Haloperidol decanoate; Behavioral: Questionnaires
- Placebo + Haloperidol (Active Comparator): Participants receive placebo, preservative free 0.9% normal saline, by vein plus a standardized dose of haloperidol 8 mg/day by vein, while in palliative care unit. Questionnaire completion at baseline, and every day while participant is in the palliative care unit. These questions will take about 20 minutes to complete
  Interventions: Drug: Placebo; Drug: Haloperidol decanoate; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Lorazepam — 3 mg by vein one time only.
  Arms: Lorazepam + Haloperidol
Drug: Placebo — Placebo consisting of preservative free 0.9% normal saline given one time by vein.
  Arms: Placebo + Haloperidol
Drug: Haloperidol decanoate — 8 mg/day by vein.
Behavioral: Questionnaires — Questionnaire completion at baseline, and every day while participant is in the palliative care unit. These questions will take about 20 minutes to complete.
  Other Names: Surveys

SUMMARY:
This randomized phase II trial studies how well haloperidol with or without lorazepam works in reducing confusion, disorientation, and inability to think or remember clearly (delirium) in patients with cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Palliative therapy with haloperidol and lorazepam may reduce symptoms of delirium and help patients with advanced cancer live more comfortably. It is not yet known whether lorazepam may be an effective treatment for delirium when given with haloperidol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the effect of single dose lorazepam and placebo as an adjuvant to haloperidol on the intensity of agitation (Richmond Agitation Sedation Scale) over 8 hours.

II. To assess the within-arm effect of single-dose lorazepam or placebo, as an adjuvant agent with haloperidol, on agitation intensity (Richmond Agitation Sedation Scale) over 8 hours in patients admitted to an acute palliative care unit.

SECONDARY OBJECTIVES:

I. To compare the effect of single dose lorazepam and placebo as an adjuvant to haloperidol on (1) delirium related distress in nurses and caregivers, (2) delirium duration, (3) need for rescue doses of neuroleptics, (4) delirium recall, (5) symptom expression (Edmonton Symptom Assessment Scale), (6) communicative capacity, (7) adverse effects, (8) discharge outcomes, and (9) survival in cancer patients.

II. To evaluate proportion of patients who consent and are randomized to study however drop out before being treated or before finishing 8-hour Richmond Agitation Sedation Scale (RASS) assessment; and the reasons of drop-outs will be documented and reported.

III. To explore the changes in biomarker levels in saliva samples (salivary cortisol, cholinesterase, C-reactive protein, interleukin-1 beta, -6, and -10) over time and in association with delirium severity.

IV. To examine the inter-rater reliability of RASS in the Acute Palliative Care Unit (APCU) setting between the bedside nurse and the research nurse at the time of study enrollment.

V. To conduct exploratory analyses on RASS as an outcome. VI. To examine the association among rescue medication use, RASS and perceived comfort by the nurses and caregivers.

VII. To examine the proportion of patients enrolled onto the delirium trial who achieved control of agitation and did not require the randomized study medication.

VIII. To identify patient factors associated with control of agitated delirium.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive lorazepam intravenously (IV) over 1-2 minutes and haloperidol IV every 6 hours or every 1 hour if needed.

ARM II: Patients receive placebo IV over 1-2 minutes and haloperidol IV every 6 hours or every 1 hour if needed.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:
* Diagnosis of advanced cancer (defined as locally advanced, metastatic, recurrent, or incurable disease)
* Admitted to Acute Palliative Care Unit (APCU)
* Delirium as per the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV- TR) criteria
* Hyperactive/mixed delirium with RASS >= 2 in the last 24 hours
* On scheduled haloperidol of =< 8 mg in the last 24 hours
* Legally authorized representative consent
* FAMILY CAREGIVERS:
* Patient's spouse, adult child, sibling, parent, other relative, or significant other (defined by the patient as a partner)
* Age 18 or older
* At the patient's bedside at least 4 hours each day during patient delirium episode
* Patients and family caregivers able to communicate in English or Spanish

Exclusion Criteria:

* PATIENTS
* History of myasthenia gravis or acute narrow angle glaucoma
* History of neuroleptic malignant syndrome
* History of Parkinson's disease or dementia
* Uncontrolled seizure disorder
* History of hypersensitivity to haloperidol or benzodiazepine
* On regular doses of benzodiazepine or chlorpromazine within the past 48 hours
* Previously documented and persistent corrected QT (QTc) prolongation (> 500 ms)
* Heart failure exacerbation at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2026-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Frisbee-Hume S, Wilson A, Dibaj SS, Nguyen T, De La Cruz M, Walker P, Zhukovsky DS, Delgado-Guay M, Vidal M, Epner D, Reddy A, Tanco K, Williams J, Hall S, Liu D, Hess K, Amin S, Breitbart W, Bruera E. Effect of Lorazepam With Haloperidol vs Haloperidol Alone on Agitated Delirium in Patients With Advanced Cancer Receiving Palliative Care: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1047-1056. doi: 10.1001/jama.2017.11468. PMID 28975307
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 1/2014 and 6/2016 from MD Anderson Cancer Center with active cancer diagnosis, having age >=18, with Delirium with Richmond Agitation-Sedation Scale score of >=2 and receiving scheduled Haloperidol 1-8 mg/day.
Pre-assignment Details: 3 patients were excluded before randomization. 1 died and 2 were ineligible.
Groups:
- Intervention Group (Lorazepam & Haloperidol): Received single dose of Lorazepam (3 mg IV, once) and Haloperidol (2mg IV, once)
- Control Group (Placebo & Haloperidol): Received single dose of Haloperidol (2mg IV, once)
Period: Overall Study
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
Started | 47 | 43
Completed | 29 | 29
Not Completed | 18 | 14
Not completed — Death | 9 | 7
Not completed — Discharged before an agitation event | 8 | 3
Not completed — Dropped out | 1 | 3
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis of 58 participants, 29 for each arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Full Range); unit: Years] | 66 [43 to 90] | 64 [30 to 88] | 65 [30 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 29 | 58
Education [Count of Participants; unit: Participants]
  High School or less | 7 | 8 | 15
  College | 11 | 6 | 17
  Completed College | 10 | 14 | 24
  Not Available | 1 | 1 | 2
Cancer Stage [Count of Participants; unit: Participants]
  Metastatic Cancer | 20 | 26 | 46
  Locally advanced | 1 | 0 | 1
  Recurrent or Persistent | 8 | 3 | 11
Cancer Type [Count of Participants; unit: Participants]
  GastroIntestinal Cancer | 9 | 4 | 13
  Hematological Cancer | 8 | 2 | 10
  Genitourinary | 2 | 1 | 3
  Head and neck | 0 | 1 | 1
  Breast | 0 | 5 | 5
  Respiratory Cancer | 4 | 10 | 14
  Gynecological | 2 | 2 | 4
  Other | 4 | 4 | 8
Karnofsky performance status [Count of Participants; unit: Participants] — The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
  Participants
    10% | 7 | 5 | 12
    20% | 15 | 12 | 27
    30% | 4 | 10 | 14
    40% | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Richmond Agitation-Sedation Scale Score (Baseline to 8 hr), Points
Description: The primary outcome was change in Richmond Agitation-Sedation Scale score from baseline to 8 hours after treatment administration. Richmond Agitation-Sedation Score ranged from -5 (unarousable) to +4 (very agitated) , where 0 denotes a calm and alert patient.
Time Frame: Baseline to 8 hours
Population: Intent to treat 58 participants, a total of 29 for each arm; 3 participants were lost to follow up from each arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
Number analyzed (Participants) | 26 | 26
score on a scale | -4.1 [-4.8 to -3.4] | -2.3 [-2.9 to -1.6]

2. Primary Outcome: Absolute Richmond Agitation-Sedation Scale Score at 8 Hour, Points
Description: Absolute score of Richmond Agitation-Sedation Scale at 8 hr, points. Richmond Agitation-Sedation Score ranged from -5 (unarousable) to +4 (very agitated) , where 0 denotes a calm and alert patient.
Time Frame: 8 hours
Population: Intent to treat 58 participants, a total of 29 for each arm; 3 participants were lost to follow up from each arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
Number analyzed (Participants) | 26 | 26
score on a scale | -2.5 [-3.2 to -1.9] | -0.7 [-1.3 to -0.1]

3. Secondary Outcome: Change in Richmond Agitation-Sedation Scale Score From Baseline to 30 Min
Description: Change in Richmond Agitation-Sedation Scale score from baseline to 30 min. Richmond Agitation-Sedation Score ranged from -5 (unarousable) to +4 (very agitated) , where 0 denotes a calm and alert patient.
Time Frame: Baseline to 30 minutes
Population: Intent to treat 58 participants, a total of 29 for each arm
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
Number analyzed (Participants) | 29 | 29
score on a scale | -3.6 [-4.3 to -2.9] | -1.6 [-2.2 to -1.0]

4. Secondary Outcome: Number of Participants With Richmond Agitation-Sedation Scale Score >=1 Within 8 hr
Description: Number of participants with Richmond Agitation-Sedation Scale score >=1 within 8 hr. Richmond Agitation-Sedation Score ranged from -5 (unarousable) to +4 (very agitated) , where 0 denotes a calm and alert patient.
Time Frame: Baseline to 8 hours
Population: Intent to treat 58 participants, a total of 29 from each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
Number analyzed (Participants) | 29 | 29
Participants | 8 | 22

ADVERSE EVENTS:
Time Frame: Baseline up to 3 days
Description: UKU (Udvalg for Kliniske Undersøgelser ) Adverse events Assessment. Total intent to treat = 58 (29+29); Total Participants used for the All Cause Mortality in both Arms, Intervention (47), and Placebo (43). The total number of deaths in the Intervention Group were 10 which includes 9 from the incomplete category and 1 from the complete category. The total number of deaths in the Control Group were 10 which includes 7 from the incomplete category and 3 from the complete category.
Arm/Group | Intervention Group (Lorazepam & Haloperidol) | Control Group (Placebo & Haloperidol)
All-Cause Mortality (participants affected / at risk) | 10/47 | 10/43
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 3/29 | 4/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Lorazepam & Haloperidol) (N=29) | Control Group (Placebo & Haloperidol) (N=29)
Hypokinesia (Musculoskeletal and connective tissue disorders) | 3 | 4
Hyperkinesia (Musculoskeletal and connective tissue disorders) | 1 | 2
Akathisia (Musculoskeletal and connective tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes